CLINICAL TRIAL: NCT02406950
Title: Preventive Effects of Sitagliptin on Endothelial Dysfunction Induced by Forearm Ischemia-Reperfusion Injury Model
Brief Title: Sitagliptin and Endothelial Dysfunction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Weon Kim, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Signal
Record Dates: First submitted 2015-03-14; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Sitagliptin; Endothelium; Ischemia-Reperfusion Injury; human
MeSH Terms: conditions — Reperfusion Injury | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitagliptin (Experimental): All participant will exam brachial artery endothelium-dependent flow-mediated dilatation (FMD). After then, pneumatic cuff wiil be inflated to 200 mmHg for 15 minutes to induce brachial artery ischemia. At the end of ischemia, 15 minutes of reperfusion was performed to induce reperfusion injury. After ischemia-reperfusion (IR) injury, brachial artery FMD will be measured again. After randomization, sitagliptin group will be treated by single dose of sitagliptin (Januvia) 50mg. In 2 hours later, brachial artery FMD measurement, IR injury and brachial artery FMD measurement will be measured again.
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): After brachial artery FMD measurement, IR injury for each 15 minutes will be performed, and brachial artery FMD will be measured again. After randomization, placebo group will be treated by nothing. In 2 hours later, brachial artery FMD measurement, IR injury and brachial artery FMD measurement will be measured again.
- Sitagliptin and glibenclimide (Other): If sitagliptin treatment show preventive effects of IR injury, the investigator will perform additional experiment to explore the mechanism (Protocol 2 study). Additional 15 healthy volunteers will be treated 5 mg of glibenclamide (Euglucon) 1 hour before administration of 50 m g of sitagliptin. In 2 hours after sitagliptin administration, FMD measurement before and after IR injury will be performed as described above.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — The brachial FMD before and after IR injury will be assessed. After randomization, study medication will be treated. In 2 hours later, the brachial FMD before and after IR injury will be assessed again. All volunteers had a wash-out period of 7 days. Seven days later, the subjects returned to crossover study medication (ie, sitagliptin or placebo), and the protocol described above was repeated.
  Other Names: Januvia
  Arms: Sitagliptin; Sitagliptin and glibenclimide

SUMMARY:
Over the years, numbers of cardioprotective drugs have been evaluated to attenuate lethal ischemia-reperfusion (IR) injuries. There is little study whether sitagliptin protects against endothelial dysfunction induced by IR injury in humans.

DETAILED DESCRIPTION:
Glucagon-like peptide-1 (GLP-1) is a novel insulinotropic peptide which is rapidly degraded by the enzyme dipeptidyl peptidase-4 (DPP-4). In addition to its attractive merit in type 2 diabetes, interest in the cardioprotective effects of GLP-1 has been increased with various reports and evidence. Previously, the investigators could show exenatide, GLP-1 receptor agonist protects ischemic/reperfusion injury-induced endothelial dysfunction through opening of KATP (ATP-sensitive potassium) channels in human ischemic/reperfusion injury model. But, recent clinical studies showed 2 different DPP-4 inhibitors, alogliptin and saxagliptin, did not decrease major adverse cardiovascular events even though improving glycemic control. The investigators will investigate the role of sitagliptin in human ischemic/reperfusion (IR) injury model of forearm conductance vessels as previous described method.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer age 20 to 40 years
* non-smoker

Exclusion Criteria:

* High blood pressure (>140/90 mmHg) or any antihypertensive medications
* diabetes
* any cardiovascular disease
* kidney disease
* thyroid disease
* cerebrovascular disease
* liver disease (bilirubin level >2 mg/dl)
* pregnancy
* body mass index >25 kg/m2

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The difference of FMD [brachial artery endothelium-dependent flow-mediated dilatation] after IR injury (brachial FMD before and after IR injury will be assessed) | 2 hours after study drug treatment

SECONDARY OUTCOMES:
The difference of FMD after IR injury in co-treatment of glibenclimide and sitagliptin ((brachial FMD before and after IR injury will be assessed) | 3.5 hours after study drug treatment

OTHER OUTCOMES:
Adverse events | 3 weeks
  Adverse events such as hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, MD, PhD, Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Kyung Hee University Hospital, Seoul, Seoul, South Korea